CLINICAL TRIAL: NCT02774928
Title: Clinical Profile of Patients With Pulmonary Hypertension Due to Lung Diseases ( Single Center Experience)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Elshazly, Professor of pulmonary Medicine, Cairo University
Other Study IDs: Cairo2001
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; COPD; ILD; OSA
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Chronic Obstructive Pulmonary Disease: Chronic Obstructive Pulmonary Disease (COPD) is a major cause of morbidity and mortality throughout the world.COPD, a common preventable and treatable disease, is characterized by persistent airflow limitation that is usually progressive and associated with an enhanced chronic inflammatory response in the airways and the lung to noxious particles or gases. Exacerbations and comorbidities contribute to the overall severity in individual patients.Spirometry is required to make a clinical diagnosis of COPD; the presence of a post-bronchodilator FEV1/FVC < 0.70 confirms the presence of persistent airflow limitation and thus of COPD .
- Interstitial lung diseases: Interstitial lung disease is a general category that includes many different lung conditions. All interstitial lung diseases affect the interstitium, a part of the lungs' anatomic structure.
- Obstructive sleep apnea (OSA): Obstructive sleep apnea (OSA) is a sleep disorder that involves cessation or significant decrease in airflow in the presence of breathing effort. It is the most common type of sleep-disordered breathing and is characterized by recurrent episodes of upper airway collapse during sleep.
  These episodes are associated with recurrent oxyhemoglobin desaturations and arousals from sleep.
  OSA that is associated with excessive daytime sleepiness is commonly called obstructive sleep apnea syndrome-also referred to as obstructive sleep apnea-hypopnea syndrome.

SUMMARY:
Development of pulmonary hypertension (PH) in chronic lung diseases has both functional and prognostic implications .

PH in Lung diseases is usually mild to moderate with preserved cardiac output, and evolves slowly alongside the progression of lung disease and hypoxemia .

However, a minority of patients develop severe PH with elevations in pulmonary artery pressure that have been described as ''out of proportion'' to the underlying disease .

The aim of this study is to compare the characteristics and outcomes of consecutive patients with PH-due to lung diseases diagnosed at our specialist referral center over a 1-year period.

DETAILED DESCRIPTION:
Development of pulmonary hypertension (PH) in chronic lung diseases has both functional and prognostic implications .

PH in Lung diseases is usually mild to moderate with preserved cardiac output, and evolves slowly alongside the progression of lung disease and hypoxemia .

However, a minority of patients develop severe PH with elevations in pulmonary artery pressure that have been described as ''out of proportion'' to the underlying disease .

Hypotheses for the etiology of this phenotype include greater susceptibility to alveolar hypoxia and/or tobacco smoke , destruction of the capillary vascular bed , inflammatory factors initiating remodeling of the pulmonary vascular bed or the coexistence of idiopathic pulmonary arterial hypertension (IPAH) in patients with lung disease .

Severe PH-lung disease has been arbitrarily defined by a resting mean pulmonary artery pressure (PAP) ≥35 mmHg by RHC . The high and increasing prevalence of chronic lung diseases and the substantial consequences of developing severe PH have generated increasing interest in PH-lung diseases.

Pulmonary vascular research unit at Chest department at Kasr-Alani school of Medicine delivers regional, adult PH service to a population with a chronic lung disease.

The aim of this study is to compare the characteristics and outcomes of consecutive patients with PH-due to lung diseases diagnosed at our specialist referral center over a 1-year period.

Patients diagnosed as chronic lung diseases( COPD,ILD,OSA,Sarcoidosis) will be recruited from out-patient's clinics & inpatients wards of Internal medicine & Chest departments, Kasr Al-ainy hospital (from June 2016 to May 2015) A written informed consent matching with Helsinki declaration will be taken from all patients.

2.2 Study methods:

All the enrolled patients will go through the following basically:

1. Detailed standard Demographic & clinical parameters.
2. Assessment of exercise tolerance (6 MWD & WHO functional capacity)
3. Assessment of pulmonary function by PFTs.
4. ECG: (Right ventricular strain,Right axis deviation,Right bundle branch block,& Left side changes 0
5. Echocardiographic evaluation for PAH: ( Right atrial area ,Right ventricular area ,Tricuspid regurgitant jet velocity (TR) ,Tricuspid annular plane systolic excursion)
6. Radiography: including chest X-ray, HRCT chest, V/Q scan& CT angiography if needed

10. RT sided heart catheterization:

* mPAP
* PCWP
* PVR
* CARDIAC INDEX 11. Statistical analysis: ……..

The subjects will be classified according to RHC into either

* Non PAH groups mPAP ≤ 21mmHG
* PAH mPAP≥ 25 mmHG:

  * Severe PH-lung diseases mPAP ≥ 35 mmgh

ELIGIBILITY:
Inclusion Criteria:

1. COPD diagnosed according to Gold 2015
2. Interstial lung diseases
3. Obstructive Sleep Apnea
4. sarcoidosis

Exclusion Criteria:

* Bronchogenic carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic lung diseases COPD ILD OSA sarcodosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
prevalence of PH | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa I Elshazly, MD, Principal Investigator — Kasr Alaini school of Medicine; Yusif Amin, MD, Study Director — Kasr Alaini school of Medicine
Locations (1):
- Kasr Alaini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
publication at international journal